CLINICAL TRIAL: NCT06912516
Title: PULSE OXIMETRY Performance Test for Vitacam. Controlled Desaturation Test.
Brief Title: PULSE OXIMETRY Performance Test for a Software Medical Device 'Vitacam'
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vitacam (Industry)
Collaborators: Tampere University (Other); Tampere University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: R23022L
Record Dates: First submitted 2025-03-25; First posted 2025-04-04 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-03

CONDITIONS: Pulse Oximetry
Keywords: Oxygen saturation; remote photoplethysmography; pulse oximetry

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Desaturation subjects (Other): This is a single arm study where healthy volunteers were subjected to a controlled desaturation protocol to ascertain if the investigational device could correctly track changes in oxygen saturation.
  Interventions: Procedure: Controlled desaturation

INTERVENTIONS:
Procedure: Controlled desaturation — A subject rests comfortably on a hospital bed, so that they do not have to move during the desaturation process.
  The subject wears the altitude simulator head bivy and breathes freely without any oxygen regulation. During the measurement, the time in low O2 saturation plateaus is limited to ten minutes in each desaturation plateau.
  They are monitored with ECG, clinical pulse oximeter, EtCO2 from non-invasive capnography with nasal cannulas and periodically non-invasive blood pressure. The monitoring is supervised by two medical doctors, present during the entire duration of the study.

SUMMARY:
This clinical investigation aims to collect data for algorithm development and testing of Vitacam as well as to later validate the system using a simultaneously collected, but segregated, hold-out validation dataset. Vitacam is a software medical device for measuring vital signs, manufactured by NE Device SW Oy. It analyses digital video recorded using a smart device with a camera to locate a subject's face and chest region. From both these regions of interest, the video is further analysed to obtain the heart rate, heartbeat intervals, respiratory rate and oxygen saturation. These measurements are used as inputs to clinical decision making. Vitacam uses remote photoplethysmography to obtain the heart rate and heartbeat intervals, and will build on this to obtain oxygen saturation using information from red-green-blue channels.

The main focus of this study is to validate the oxygen saturation, heart rate and heartbeat intervals measured by Vitacam against gold standard references, applying the ISO 80601:2019 standard.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-40 years
* ASA category 1
* Positive Allen's test
* Passing the physical examination
* Ability to give informed consent
* Volunteering for the study
* Fluent Finnish or English

Exclusion Criteria:

* Age under 18 years or over 40 years
* Smoker
* Pregnancy
* Does not pass the physical examination
* Negative Allen's test
* Relevant medical illnesses
* Cardiovascular disease
* Pulmonary disease
* Inability to give informed consent
* Denial

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2023-12-22 (Actual); Primary Completion 2024-09-15 (Actual); Study Completion 2024-11-01 (Actual)

PRIMARY OUTCOMES:
Accuracy of oxygen saturation measurements - Root Mean Square Error | A 30-45 minute period during which the participant is subjected to the de-saturation process
  Accuracy as measured by Root Mean Square Error should be less than or equal to 4% for SpO2 as per ISO 80601-2-61:2019. It is calculated from the difference of the SpO2 measured from the investigational device and that of the reference device.
Accuracy of oxygen saturation measurements - Mean absolute error | A 30-45 minute period during which the participant is subjected to the de-saturation process
  Accuracy as measured by Mean Absolute Error should be less than or equal to 4% for SpO2 as per ISO 80601-2-61:2019. It is calculated from the difference of the SpO2 measured from the investigational device and that of the reference device.

SECONDARY OUTCOMES:
Accuracy of interbeat intervals of the investigational device against successive R waves of the QRS complex from an Electrocardiogram | A 30-45 minute period during which the participant is subjected to the de-saturation process
  To validate the accuracy of Vitacam interbeat intervals, both the intervals and heart rate variability metrics derived from these intervals, will be compared to the RR intervals and heart rate variability metrics derived from a 5-lead ECG

CONTACTS AND LOCATIONS:
Locations (1):
- Tampere University, Tampere, Finland, Finland

IPD SHARING:
Plan to Share IPD: No
IPD cannot be shared due to GDPR